CLINICAL TRIAL: NCT03075644
Title: A Multicentre, Randomised, Open-labelled, Parallel-group, Activecontrolled Trial to Evaluate the Safety of Once Weekly Dosing of Somapacitan (NNC0195-0092) and Daily Norditropin® FlexPro® for 52 Weeks in Previously Human Growth Hormone Treated Japanese Adults With Growth Hormone Deficiency
Brief Title: A Trial to Evaluate the Safety of Once Weekly Dosing of Somapacitan (NNC0195-0092) and Daily Norditropin® FlexPro® for 52 Weeks in Previously Human Growth Hormone Treated Japanese Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN8640-4244; U1111-1181-1618 (Other: World Health Organization (WHO)); JapicCTI-173534 (Registry Identifier: JAPIC)
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Growth Hormone Disorder; Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somapacitan (Experimental)
  Interventions: Drug: somapacitan
- Norditropin (Active Comparator)
  Interventions: Drug: Norditropin

INTERVENTIONS:
Drug: somapacitan — Once weekly subcutaneous injections (s.c., under the skin)
  Arms: Somapacitan
Drug: Norditropin — Daily subcutaneous injections (s.c., under the skin)
  Arms: Norditropin

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate the safety of once weekly dosing of somapacitan (NNC0195-0092) and daily Norditropin® FlexPro® for 52 weeks in previously human growth hormone treated Japanese adults with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria: - Male or female of at least 18 years of age and not more than 79 years of age at the time of signing informed consent - GHD diagnosed for at least 6 months (defined as 180 days) prior to screening - Treatment with hGH for at least 6 consecutive months (defined as 180 days) at screening - If applicable, hormone replacement therapies for any other hormone deficiencies, adequate and stable for at least 90 days prior to randomisation as judged by the investigator Exclusion Criteria: - Active malignant disease or history of malignancy. Exceptions to this exclusion criterion:1/ Resected in situ carcinoma of the cervix and squamous cell or basal cell carcinoma of the skin with complete local excision 2/ Subjects with GHD attributed to treatment of intracranial malignant tumours or leukaemia, provided that a recurrence-free survival period of at least 5 years is documented in the subject's medical records - For subjects with surgical removal or debulking of pituitary adenoma or other benign intracranial tumour within the last 5 years:Evidence of growth of pituitary adenoma or other benign intracranial tumour within the last 12 months (defined as below or equal to 365 days) before randomisation. Absence of growth must be documented by two post-surgery magnetic resonance imaging (MRI) scans or CT scans. The most recent MRI or CT scan must be performed below or equal to 9 months (defined as below or equal to 270 days) prior to randomisation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Japan (12):
  - Novo Nordisk Investigational Site, Bunkyo-ku, Tokyo
  - Novo Nordisk Investigational Site, Chiba-shi, Chiba
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Kagoshima
  - Novo Nordisk Investigational Site, Kobe, Hyogo
  - Novo Nordisk Investigational Site, Kyoto-shi Kyoto
  - Novo Nordisk Investigational Site, Okayama, Okayama
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Sagamihara-shi, Kanagawa
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Yamagata-shi, Yamagata
  - Novo Nordisk Investigational Site, Yokohama, Kanagawa

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Otsuka F, Takahashi Y, Tahara S, Ogawa Y, Hojby Rasmussen M, Takano K. Similar safety and efficacy in previously treated adults with growth hormone deficiency randomized to once-weekly somapacitan or daily growth hormone. Clin Endocrinol (Oxf). 2020 Nov;93(5):620-628. doi: 10.1111/cen.14273. Epub 2020 Aug 14. PMID 32603494
- [Derived] Takahashi Y, Biller BMK, Fukuoka H, Ho KKY, Rasmussen MH, Nedjatian N, Svaerke C, Yuen KCJ, Johannsson G. Weekly somapacitan had no adverse effects on glucose metabolism in adults with growth hormone deficiency. Pituitary. 2023 Feb;26(1):57-72. doi: 10.1007/s11102-022-01283-3. Epub 2022 Nov 15. PMID 36380045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 12 sites in Japan.
Pre-assignment Details: Participants were randomised in a 3:1 manner to receive either somapacitan or Norditropin®.
Groups:
- Norditropin®: Participants were to receive a subcutaneous (s.c.) injection of Norditropin® once daily for 52 weeks (20 weeks of dose titration and 32 weeks of fixed dose treatment). The dose was titrated every fourth week starting from week 4 based on insulin like growth factor-I standard deviation score (IGF-I SDS) values. The starting dose was 0.2 milligrams per day (mg/day) for participants between 18 and 60 years of age; 0.3 mg/day for females on oral oestrogen irrespective of age; and 0.1 mg/day for participants older than 60 years. The maximum daily dose of Norditropin® was 1.0 milligram (mg).
- Somapacitan: Participants were to receive a s.c. injection of somapacitan once weekly for 52 weeks (20 weeks of dose titration and 32 weeks of fixed dose treatment). The dose was titrated every fourth week starting from week 4 based on IGF-I SDS values. The starting dose was 1.5 milligrams per week (mg/week) for participants between 18 and 60 years of age; 2.0 mg/week for females on oral oestrogen irrespective of age; and 1.0 mg/week for participants older than 60 years. The maximum weekly dose of somapacitan was 8 mg.
Period: Overall Study
Arm/Group | Norditropin® | Somapacitan
Started | 16 | 46
Full Analysis Set (FAS) | 16 | 46
Safety Analysis Set (SAS) | 16 | 46
Completed | 15 | 45
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised participants that received at least one dose of randomised treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Norditropin® | Somapacitan | Total
Number analyzed (Participants) | 16 | 46 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.3 (11.5) | 54.1 (12.1) | 52.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 22 | 29
  Male | 9 | 24 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 46 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 46 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events, Including Injection Site Reactions
Description: An adverse event (AE) was any untoward medical occurrence in a participant administered a medicinal product, and which did not necessarily have a causal relationship with the treatment. Rate of AEs per 100 patient years at risk with onset after the first administration of trial product and up until end of the trial (53 weeks) or 14 days after last trial drug administration, whichever came first, are presented.
Time Frame: Weeks 0-53
Population: Safety analysis set (SAS) which comprised all randomised participants who received at least one dose of randomised treatment.
Measure: Number; unit: Event rate per 100 patient years
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
Event rate per 100 patient years | 309.8 | 312.7

2. Secondary Outcome: Change in Cross-sectional Total Adipose Tissue Compartments
Description: Cross-sectional total adipose tissue compartments (TAT) were determined by quantitative computed tomography (CT) scans. Change from baseline (week 0) to end of treatment period (52 weeks) in cross-sectional TAT compartments is presented.
Time Frame: Week 0, week 52
Population: FAS comprised all randomised participants who received at least one dose of randomised treatment. Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Square centimeters (cm^2)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 43
Square centimeters (cm^2) | 7.450 (32.177) | -7.091 (58.893)

3. Secondary Outcome: Change in Subcutaneous Adipose Tissue Compartments
Description: Subcutaneous adipose tissue compartments (SAT) was determined by quantitative CT scans. Change from baseline (week 0) to end of treatment period (52 weeks) in SAT compartments is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 43
cm^2 | 6.779 (22.900) | -5.033 (40.735)

4. Secondary Outcome: Change in Intra-abdominal or Visceral Adipose Tissue Compartments
Description: Intra-abdominal or visceral adipose tissue (VAT) compartments was determined by quantitative CT scans. Change from baseline (week 0) to end of treatment period (52 weeks) in VAT compartments is presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
cm^2 | 0.671 (15.284) | -2.618 (29.123)

5. Secondary Outcome: Change in Treatment Satisfaction Questionnaire for Medication (TSQM-9) Scores
Description: The Treatment Satisfaction Questionnaire for Medication - 9 items (TSQM-9) is a generic questionnaire that measures a patients' satisfaction with medication. Items are rated on a 5-point or 7-point scale according to patients' experience with the medication. The items covered are satisfaction with the effectiveness of the medication, convenience and global satisfaction of treatment. Each domain is based on 3 questions. The score is calculated in a range from 0 to 100, where a higher score reflects a better outcome. Scores have been summed and then scaled to 0-100. Change in TSQM-9 scores from baseline (week 0) to week 52 are presented.
Time Frame: Week 0, week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Score on a scale
  Effectiveness | 3.6 (16.2) | 7.9 (17.5)
  Convenience | 8.7 (9.9) | 13.3 (17.3)
  Global satisfaction | 3.1 (11.1) | 10.0 (16.8)

6. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters were evaluated for head, ears, eyes, nose, throat, neck; respiratory system; cardiovascular system, gastrointestinal system, incl. mouth; musculoskeletal system; nervous system (central and peripheral); skin; and lymph node palpation. The investigator evaluated the findings from the physical examination and classifies them as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS). Results are presented for week 0 and week 52.
Time Frame: Week 0, week 52
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of randomised treatment. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
Participants
  Week 0: Head, ears, eyes, nose, throat, neck: Normal | 15 | 45
  Week 0: Head, ears, eyes, nose, throat, neck: Abnormal NCS | 0 | 1
  Week 0: Head, ears, eyes, nose, throat, neck: Abnormal CS | 1 | 0
  Week 52: Head, ears, eyes, nose, throat, neck: number analyzed (Participants) | 15 | 45
  Week 52: Head, ears, eyes, nose, throat, neck: Normal | 14 | 43
  Week 52: Head, ears, eyes, nose, throat, neck: Abnormal NCS | 0 | 1
  Week 52: Head, ears, eyes, nose, throat, neck: Abnormal CS | 1 | 1
  Week 0: Respiratory system: Normal | 16 | 46
  Week 0: Respiratory system: Abnormal NCS | 0 | 0
  Week 0: Respiratory system: Abnormal CS | 0 | 0
  Week 52: Respiratory system: number analyzed (Participants) | 15 | 45
  Week 52: Respiratory system: Normal | 15 | 45
  Week 52: Respiratory system: Abnormal NCS | 0 | 0
  Week 52: Respiratory system: Abnormal CS | 0 | 0
  Week 0: Cardiovascular system: Normal | 16 | 46
  Week 0: Cardiovascular system: Abnormal NCS | 0 | 0
  Week 0: Cardiovascular system: Abnormal CS | 0 | 0
  Week 52: Cardiovascular system: number analyzed (Participants) | 15 | 45
  Week 52: Cardiovascular system: Normal | 15 | 44
  Week 52: Cardiovascular system: Abnormal NCS | 0 | 1
  Week 52: Cardiovascular system: Abnormal CS | 0 | 0
  Week 0: Gastrointestinal system: Normal | 15 | 46
  Week 0: Gastrointestinal system: Abnormal NCS | 1 | 0
  Week 0: Gastrointestinal system: Abnormal CS | 0 | 0
  Week 52: Gastrointestinal system: number analyzed (Participants) | 15 | 45
  Week 52: Gastrointestinal system: Normal | 15 | 45
  Week 52: Gastrointestinal system: Abnormal NCS | 0 | 0
  Week 52: Gastrointestinal system: Abnormal CS | 0 | 0
  Week 0: Musculoskeletal system: Normal | 16 | 45
  Week 0: Musculoskeletal system: Abnormal NCS | 0 | 1
  Week 0: Musculoskeletal system: Abnormal CS | 0 | 0
  Week 52: Musculoskeletal system: number analyzed (Participants) | 15 | 45
  Week 52: Musculoskeletal system: Normal | 15 | 43
  Week 52: Musculoskeletal system: Abnormal NCS | 0 | 0
  Week 52: Musculoskeletal system: Abnormal CS | 0 | 2
  Week 0: Nervous system: Normal | 16 | 46
  Week 0: Nervous system: Abnormal NCS | 0 | 0
  Week 0: Nervous system: Abnormal CS | 0 | 0
  Week 52: Nervous system: number analyzed (Participants) | 15 | 45
  Week 52: Nervous system: Normal | 15 | 45
  Week 52: Nervous system: Abnormal NCS | 0 | 0
  Week 52: Nervous system: Abnormal CS | 0 | 0
  Week 0: Skin: Normal | 16 | 46
  Week 0: Skin: Abnormal NCS | 0 | 0
  Week 0: Skin: Abnormal CS | 0 | 0
  Week 52: Skin: number analyzed (Participants) | 15 | 45
  Week 52: Skin: Normal | 15 | 44
  Week 52: Skin: Abnormal NCS | 0 | 1
  Week 52: Skin: Abnormal CS | 0 | 0
  Week 0: Lymph node palpation: Normal | 16 | 44
  Week 0: Lymph node palpation: Abnormal NCS | 0 | 2
  Week 0: Lymph node palpation: Abnormal CS | 0 | 0
  Week 52: Lymph node palpation: number analyzed (Participants) | 15 | 45
  Week 52: Lymph node palpation: Normal | 15 | 45
  Week 52: Lymph node palpation: Abnormal NCS | 0 | 0
  Week 52: Lymph node palpation: Abnormal CS | 0 | 0

7. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week -3) in body weight at week 52 is presented.
Time Frame: Week -3, week 52
Population: SAS comprised all randomised participants who received at least one dose of randomised treatment. Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (Kg)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Kilogram (Kg) | 0.66 (2.50) | -0.29 (3.49)

8. Secondary Outcome: Change in SBP and DBP
Description: Change from baseline (week 0) in systolic blood pressure (SBP) and diastolic blood pressure (DBP) at week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Millimeters of mercury (mmHg)
  SBP | -3.1 (14.8) | -3.3 (11.7)
  DBP | 1.1 (9.7) | 0.9 (8.7)

9. Secondary Outcome: Change in Pulse
Description: Change from baseline (week 0) in pulse at week 52 is presented.
Time Frame: Week 0, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Beats per minute | -1.1 (7.5) | 1.4 (8.9)

10. Secondary Outcome: Change in ECG
Description: The ECG was assessed by the investigator at baseline (week -3) and week 52 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at week -3 and week 52 are presented.
Time Frame: Week -3, week 52
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
Participants
  week -3: Normal | 16 | 39
  week -3: Abnormal NCS | 0 | 7
  week -3: Abnormal CS | 0 | 0
  week 52: number analyzed (Participants) | 15 | 45
  week 52: Normal | 15 | 37
  week 52: Abnormal NCS | 0 | 8
  week 52: Abnormal CS | 0 | 0

11. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change from baseline (week -3) in haemoglobin at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Grams/liter (g/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Grams/liter (g/L) | -2.071 (7.790) | 0.311 (6.026)

12. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change from baseline (week -3) in haematocrit at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage point of haematocrit
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Percentage point of haematocrit | -0.64 (2.76) | 0.04 (2.31)

13. Secondary Outcome: Change in Haematology: Thrombocytes, Leucocytes
Description: Change from baseline (week -3) in thrombocytes and leucocytes at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
10^9 cells/L
  Thrombocytes: number analyzed (Participants) | 14 | 44
  Thrombocytes | 0.1 (27.7) | 5.7 (33.5)
  Leucocytes: number analyzed (Participants) | 14 | 45
  Leucocytes | -0.29 (1.01) | -0.50 (1.43)

14. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change from baseline (week -3) in erythrocytes at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cells per picoliter
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
cells per picoliter | -0.086 (0.271) | -0.007 (0.228)

15. Secondary Outcome: Change in Haematology: Mean Corpuscular Volume
Description: Change from baseline (week -3) in mean corpuscular volume at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Femtoliters (fL)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Femtoliters (fL) | 0.00 (2.45) | 0.29 (1.91)

16. Secondary Outcome: Change in Haematology: Mean Corpuscular Haemoglobin Concentration
Description: Change from baseline (week -3) in mean corpuscular haemoglobin concentration at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Millimoles per liter (mmol/L) | 0.04 (0.47) | 0.05 (0.45)

17. Secondary Outcome: Change in Biochemistry: Creatinine, Uric Acid, and Bilirubin (Total)
Description: Change from baseline (week -3) in creatinine, uric acid, and bilirubin (total) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Micromoles per liter (umol/L)
  Creatinine | 1.4 (7.8) | 1.0 (7.4)
  Uric acid | 25.9 (41.9) | 6.7 (49.9)
  Total bilirubin | -0.21 (5.21) | 0.56 (3.81)

18. Secondary Outcome: Change in Biochemistry: Creatinine Kinase, ALT, AST, ALP and GGT
Description: Change from baseline (week -3) in creatinine kinase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and gamma-glutamyl transferase (GGT) at week 52 is presented.
Time Frame: Week -3, week 52
Population: SAS which comprised all randomised participants who received at least one dose of randomised treatment. Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Units per liter (U/L)
  Creatinine kinase | -10.4 (66.8) | 6.8 (261.3)
  ALT | -4.9 (13.4) | -1.6 (9.4)
  AST | -3.2 (10.3) | -1.4 (7.2)
  ALP | -9.1 (11.0) | -0.7 (11.4)
  GGT | -9.4 (19.2) | -0.6 (6.6)

19. Secondary Outcome: Change in Biochemistry: Urea, Sodium, Potassium, Chloride, Phosphate (Inorganic), Calcium (Total)
Description: Change from baseline (week -3) in urea, sodium, potassium, chloride, phosphate (inorganic), calcium (total) (mmol/L) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
mmol/L
  Urea | 0.29 (0.83) | 0.71 (1.29)
  Sodium | -0.3 (1.9) | 0.2 (2.8)
  Potassium | -0.04 (0.29) | 0.04 (0.34)
  Chloride | 0.4 (2.8) | 0.6 (2.9)
  Inorganic phosphate | 0.000 (0.185) | 0.028 (0.172)
  Total calcium | -0.067 (0.068) | -0.051 (0.082)

20. Secondary Outcome: Change in Biochemistry: Total Protein and Albumin
Description: Change from baseline (week -3) in total protein and albumin at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Grams/liter (g/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Grams/liter (g/L)
  Total protein | -0.6 (3.7) | 1.4 (3.1)
  Albumin | 0.3 (2.8) | 1.3 (2.4)

21. Secondary Outcome: Change in Biochemistry: eGFR Creatinine
Description: Estimated glomerular filtration rate (eGFR) creatinine (measured in milliliters per minute per 1.73 square meters [mL/min/1.73m^2]) was evaluated using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. Change from baseline (week -3) in eGFR at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
mL/min/1.73m^2 | -1.4 (7.1) | -1.4 (6.2)

22. Secondary Outcome: Change in HbA1c
Description: Change from baseline (week -3) in glycosylated haemoglobin (HbA1c) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Percentage point of HbA1c | -0.04 (0.22) | -0.07 (0.21)

23. Secondary Outcome: Change in FPG
Description: Change from baseline (week -3) in fasting plasma glucose (FPG) (mmol/L) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
mmol/L | 0.014 (0.442) | 0.089 (0.453)

24. Secondary Outcome: Change in Fasting Insulin
Description: Change from baseline (week -3) in fasting insulin at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Picomoles per liter (pmol/L) | -16.7 (54.1) | -8.7 (44.7)

25. Secondary Outcome: Change in Steady State Beta Cell Function
Description: Change from baseline (week -3) in steady state beta cell function (%B) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of beta cell function (%B)
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 12 | 39
Percentage of beta cell function (%B) | -23.58 (69.76) | -19.06 (65.61)

26. Secondary Outcome: Change in Insulin Resistance
Description: Change from baseline (week -3) in insulin resistance (IR) (Homeostatic model assessment (HOMA) estimates) at week 52 is presented.
Time Frame: Week -3, week 52
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage (%) of IR
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 14 | 45
Percentage (%) of IR | -0.60 (2.03) | -0.25 (1.70)

27. Secondary Outcome: Occurrence of Anti-somapacitan Antibodies
Description: Number of participants with anti-somapacitan antibodies at baseline (week 0) and week 53 are presented. This outcome measure is applicable only for the treatment arm "Somapacitan".
Time Frame: Weeks 0 - 53
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Somapacitan
Number analyzed (Participants) | 46
Participants
  Week 0 | 0
  Week 53 | 0

28. Secondary Outcome: Occurrence of Anti-hGH Antibodies
Description: Number of participants with anti-human growth hormone (hGH) antibodies at baseline (week 0) and week 53 are presented.
Time Frame: Weeks 0 - 53
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
Participants
  Week 0 | 0 | 1
  Week 53: number analyzed (Participants) | 15 | 46
  Week 53 | 0 | 0

29. Secondary Outcome: Incidence of Clinical Technical Complaints
Description: A technical complaint was any written, electronic, or oral communication that alleged product (medicine or device) defects. Number of partipants who reported technical complaints during the course of the trial are presented.
Time Frame: Weeks 0 - 53
Population: Overall number of participants analyzed = SAS which comprised all randomised participants who received at least one dose of randomised treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Norditropin® | Somapacitan
Number analyzed (Participants) | 16 | 46
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Weeks 0 - 53
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 14 days after the last day of trial product administration. Results are based on the SAS which comprised all randomised participants who received at least one dose of randomised treatment.
Arm/Group | Norditropin® | Somapacitan
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/16 | 4/46
Other Adverse Events (participants affected / at risk) | 11/16 | 33/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin® (N=16) | Somapacitan (N=46)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Norditropin® (N=16) | Somapacitan (N=46)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 1 (2) | 4 (4)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (3)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Injection site haemorrhage (General disorders) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (9) | 22 (46)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/44/NCT03075644/Prot_SAP_000.pdf